CLINICAL TRIAL: NCT02279576
Title: Phase II Study With Pazopanib and Weekly Paclitaxel in Metastatic or Locally Advanced Squamous Penile Carcinoma Patients Previously Treated With Cisplatin Based Chemotherapy
Brief Title: Study With Pazopanib and Weekly Paclitaxel in Penile Carcinoma (PAZOPEN-SOGUG)
Acronym: PAZOPEN-SOGUG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The low recruitment of patients will not allow to complete the study with the required number of patients within reasonable time.
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOG-CPE-2014-03; 2014-003127-22 (EudraCT Number)
Record Dates: First submitted 2014-10-27; First posted 2014-10-31 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2015-11

CONDITIONS: Penile Squamous Cell Carcinoma Stage IV
Keywords: Penile squamous cell carcinoma; Pazopanib; Weekly paclitaxel
MeSH Terms: interventions — pazopanib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib plus weekly paclitaxel (Experimental): Pazopanib 800mg /day continuously administered plus paclitaxel 65 mg/m2 in weekly administration, 3 administrations (D1, D8 and D15) every 4 weeks period.
  Interventions: Drug: Pazopanib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pazopanib — Pazopanib 800mg/day continuously administered.
  Other Names: Daily pazopanib
Drug: Paclitaxel — Paclitaxel 65 mg/m2 in weekly administration 3 administrations (D1, D8 and D15) every 4 weeks period.
  Other Names: Weekly paclitaxel

SUMMARY:
Penile cancer is an uncommon disease, with devastating physical and psychological effects on patients. Penile carcinoma even in advanced stages is responsive to several chemotherapeutic agents. However, due to the low incidence of penile cancer, no large studies have been reported concerning chemotherapy.

Various single agents were tested for activity en penile cancer in de 70s and 80s. Response rates ranged from 10 to 27% with cisplatin, 20 to 21% with bleomycin, and 0-62% with methotrexate. These agents in combination were tested in different studies. Other chemotherapy schemes have been studied, as combination of cisplatin with 5 fluorouracil with or without taxol, and cisplatin plus irinotecan. All of them in limited phase II studies, with described higher responses rates in some of them but without results confirmation in phase III studies.

In conclusion, tested regimens so far have not been very successful in advanced stages of the disease.

Antiangiogenic therapy has been demonstrated effective in the treatment of similar cancer types as lung and head and neck, so it can be postulated that antiangiogenic therapy can be effective in the treatment of penile carcinoma. Pazopanib is a new potent oral antiangiogenic therapy.

Cytotoxic agents, such as paclitaxel, when administered at low doses and frequent intervals, may exert antiangiogenic effects, thereby enhancing anticancer activity. Recently, combination of pazopanib and paclitaxel administered in a metronomic schedule (80mg/m2 weekly 3 weeks every 4 weeks cycle) obtained a 40% response rate and an 80% of disease control in the first-line treatment of melanoma patients. Treatment was well tolerated.

As paclitaxel and antiangiogenic drugs seem a very active treatment, combination of pazopanib and paclitaxel seems a good combination to be tested in patients with penile carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >= 18 years
* Histologically confirmed diagnosis of squamous cell carcinoma of the penis
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Measurable disease criteria according to RECIST criteria (version 1.1)
* Progressive disease after treatment with cisplatin or carboplatin based chemotherapy.
* Archived tumor tissue must be provided for all subjects for biomarker analysis before and/or during treatment with investigational product.
* Adequate organ system function - Haemoglobin >= 9.0 gr/dl (5.6 mmol/L) and stable in the previous 4 weeks to start study treatment - Neutrophils >= 1.5 x 10*9/L - Platelets >= 100 x 10*9/L - Total bilirubin <= 1.5 x UNL - AST/SGOT and ALT/SGPT <= 2.5 x UNL - serum creatinine <= 1.5 mg/dL - Urine protein to creatinine ratio < 1.
* Normal coagulation tests: - Prothrombin time (PT) or international normalized ratio (INR) <= 1.2 X ULN - Activated partial thromboplastin time (aPTT) <= 1.2 X ULN 10. Are able to swallow and retain oral tablets

Exclusion Criteria:

* Prior malignancy.
* Central nervous system metastases at baseline, with the exception of those subjects who have previously-treated CNS metastases (surgery ± radiotherapy, radiosurgery, or gamma knife) and who meet both of the following criteria: a) are asymptomatic and b) have no requirement for steroids or enzyme-inducing anticonvulsants
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding.
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product.
* Corrected QT interval (QTc) > 480 ms
* History of any one or more of the following cardiovascular conditions within the past 6 months: - Cardiac angioplasty or stenting - Myocardial infarction - Unstable angina - Coronary artery bypass graft surgery - Symptomatic peripheral vascular disease - Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of >= 140 mmHg or diastolic blood pressure (DBP) of >= 90 mmHg].
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage
* Recent hemoptysis (>= 1/2 teaspoon [2.5 mL]) of red blood within 8 weeks before first dose of study drug).
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subjects safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications 14 days prior to the first dose of study drug and for the duration of the study.
* Treatment with any of the following anti-cancer therapies: - radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR - chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days prior to the first dose of Pazopanib
* Administration of any non-oncologic investigational drug within 30 days prior to receiving the first dose of study treatment
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or paclitaxel and/or excipients that contraindicates their participation.
* Previous taxane or/and antiVEGF treatment would not allow patient to participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Up to 6 months
  Evaluate response rate in terms of complete and partial response (RECIST criteria version 1.1)

SECONDARY OUTCOMES:
Clinical benefit rate | Up to 6 months
  Clinical benefit rate (complete and partial response and stable disease) evaluated according RECIST criteria version 1.1
Progression free survival | Up to 12 months
  Time from patient inclusion until progression disease (RECIST criteria version 1.1) or death from any cause, whichever came first, assessed up to 12 months
Response duration | Up to 12 months
  Time from first response to progression disease (RECIST criteria version 1.1) or death from any cause, whichever came first, assessed up to 12 months
Overall survival | Up to 18 months
  Time from patient inclusion to death assessed up to 18 months
Safety tolerability profile as measured by the number of events per patient | Up to 6 months
  Number of events per patient

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Climent, MD, Study Director — Instituto Valenciano de Oncología
Locations (8):
- Spain (8):
  - Hospital de La Santa Creu I Sant Pau, Barcelona, Barcelona
  - Institut Català D'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Regional Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital General Universitario J.M. Morales Meseguer, Murcia, Murcia
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Instituto Valenciano de Oncología, Valencia, Valencia